CLINICAL TRIAL: NCT05274685
Title: Early Renal Replacement Therapy in COVID 19 Patients With AKI Improves the Prognosis of the Disease
Brief Title: Early Renal Replacement Therapy in COVID 19 Patients With AKI Does it Improve the Outcome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mokhtar Ahmed, lecturer of anesthesia and intensive care, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: soh-Med-22-2-24
Record Dates: First submitted 2022-03-09; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Multi Organ Failure
MeSH Terms: conditions — Multiple Organ Failure | interventions — Dialysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- covid positive with acute kidney injury receiving early renal replacement (Experimental)
  Interventions: Procedure: haemodialysis
- covid positive with acute kidney injury under conservative management (Experimental)
  Interventions: Procedure: haemodialysis

INTERVENTIONS:
Procedure: haemodialysis — continuous venovenous hemodiafiltration (CVVHDF) at a prescribed dose of 30-35 mL/kg/h of effluent and with regional citrate anticoagulation

SUMMARY:
patients will be divided into two equal groups, each group including 50 adult patients with a confirmed diagnosis of covid, patients with acute kidney injury, the first group will be treated with early hemodialysis, second group will be conservative until there is an urgent need for dialysis

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years old) with confirmed severe acute respiratory syndrome coronavirus 2 infections admitted to the ICU.

Exclusion Criteria:

* •Malignancy.

  * Immuno-deficiency diseases.
  * Chronic diabetic, cardiac and hypertensive patients
  * autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
reduction of Sequential Organ Failure Assessment Score | 2 weeks
  prevention of multi-organ failure associated with covid including respiratorym circulatory, liver and renal failure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No